CLINICAL TRIAL: NCT07108491
Title: The Effects of Balance Training With Progressive Intermittent Visual Occlusions on Balance, Instability, Muscle Strength, and Functional Performance in Patients With Chronic Ankle Instability (RCT)
Brief Title: Balance Training With Progressive Intermittent Visual Occlusions in Chronic Ankle Instability(RCT)
Acronym: BTPIVO-CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Miyong Jeong, Graduate Student Researcher, Sahmyook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYU 2025-01-011-002; IRB Number (Other: SYU 2025-01-011-002)
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Ankle Injuries
Keywords: Intermittent Visual Occlusions; Balance; Muscle Strength; Functional Performance; Chronic Ankle Instability
MeSH Terms: conditions — Ankle Injuries | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Participants were divided into an experimental group and a control group. The experimental group performed balance exercises while wearing stroboscopic glasses, whereas the control group performed the same balance exercises without the glasses. Both groups trained twice a week for four weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroboscopic Balance Training Group (Experimental): The experimental group performed balance training with stroboscopic glasses twice a week for four weeks
  Interventions: Biological: Balance Training with Stroboscopic Glasses
- Control Group (General Balance Training) (Active Comparator): The control group performed the same balance training twice a week for four weeks
  Interventions: Biological: Balance Training without Glasses

INTERVENTIONS:
Biological: Balance Training with Stroboscopic Glasses — The difficulty level of intermittent visual occlusion was structured from Level 1 to Level 8 based on frequency. As the flicker speed of the lenses decreased and the frequency lowered, the difficulty increased. For example, a setting of 6 Hz means the lenses flicker six times per second, whereas 1 Hz indicates one flicker per second.
  Levels 1 to 5 are suitable for dynamic movements such as catching or hitting a ball, while Levels 3 to 8 are appropriate for balance and proprioceptive training.
  In this study, participants wore stroboscopic glasses (Senaptec Strobe, Senaptec, USA, 2016) and began at Level 1 (6 Hz). The difficulty was gradually increased each week, with the setting adjusted to Level 3 (4 Hz) in Week 2, Level 4 (3 Hz) in Week 3, and Level 5 (2.25 Hz) in Week 4 (see Table 5).
  The training was conducted using the standard Mode A, in which both lenses flicker simultaneously.
  Arms: Stroboscopic Balance Training Group
Biological: Balance Training without Glasses — The exercise program consisted of six types of exercises and was conducted in a 30-minute circuit training format repeated twice per session. Participants took part in two sessions per week for four weeks, totaling eight sessions. The six exercises were completed as a circuit, repeated twice per session. A 30-second rest was provided between exercises and a 2-minute rest between circuits. All exercises were conducted by a licensed physical therapist to ensure safety.
  Arms: Control Group (General Balance Training)

SUMMARY:
Based on the purpose of this study, the following hypotheses were established:

There will be a significant difference in balance changes within and between groups following balance training with progressive intermittent visual occlusions compared to general balance training.

There will be a significant difference in instability changes within and between groups following balance training with progressive intermittent visual occlusions compared to general balance training.

There will be a significant difference in muscle strength changes within and between groups following balance training with progressive intermittent visual occlusions compared to general balance training.

There will be a significant difference in functional performance changes within and between groups following balance training with progressive intermittent visual occlusions compared to general balance training.

DETAILED DESCRIPTION:
In this study, participants were voluntarily recruited through social networking services, university bulletin boards, and in-hospital advertisements at N Hospital in Seoul. A total of 28 participants were provided with sufficient information regarding the purpose, procedures, and assessment methods of the study. After obtaining written informed consent, the participants were randomly assigned into either the experimental group (n = 14), which received balance training with progressive intermittent visual occlusions, or the control group (n = 14), which received general balance training only, using the randomization website (www.randomizer.org). Random assignment was conducted in a single-blind manner, and participants were unaware of their group allocation.

During the pre-intervention assessment, general characteristics (sex, side tested, age, height, weight, BMI, leg length) were recorded. Measures of balance, instability, muscle strength, and functional performance were taken. Each variable was measured three times to reduce error, and the average value was calculated.

Interventions were conducted individually in a designated private space, and participants were scheduled according to their availability. The experimental group participated in balance training with progressive intermittent visual occlusions twice a week for four weeks (eight sessions in total), with each session lasting 30 minutes. The control group performed the same balance training protocol without wearing stroboscopic glasses.

All interventions were administered by an experienced physical therapist with more than 10 years of clinical experience. Pre- and post-assessments were conducted by a blinded assessor who was unaware of the participants' group allocation. All procedures before and after the intervention were conducted under the same conditions. Following the intervention, balance, instability, muscle strength, and functional performance were reassessed using the same protocols as in the pretest.

During the intervention period, one participant in the experimental group dropped out due to plantar foot pain, resulting in a final sample size of 13 in the experimental group and 14 in the control group for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria

History of recurrent ankle sprains within the 12 months prior to the study

At least two episodes of the ankle "giving way"

Current ankle instability, indicated by a Cumberland Ankle Instability Tool (CAIT) score of 24 or less

Exclusion Criteria

History of lower extremity fracture or musculoskeletal surgery

Lower extremity injury within the past 3 months

Vestibular disorders or uncorrectable visual impairments

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
dynamic balance | At baseline (pre-intervention) and 4 weeks after completing the intervention
  Dynamic balance ability was assessed using the Y-Balance Test. The posterior-medial and posterior-lateral directions were set at 90 degrees to each other, and each was set at 135 degrees relative to the anterior direction. The directions were determined based on the supporting leg. Participants performed three practice trials followed by three test trials for each direction. All measurements were conducted barefoot, and reach distances were measured in centimeters using a measuring tape. Participants stood at the center point where the tape lines intersected and reached as far as possible in the anterior, posterior-medial, and posterior-lateral directions.
Static balance | At baseline (pre-intervention) and 4 weeks after completing the intervention
  Static balance ability was assessed using the Modified Static Postural Stability Test. Participants stood on one leg with the knee fully extended and maintained a heel-raised position, lifting the heel approximately 2-3 cm off the ground. The measurement was stopped if balance was lost, and the duration of maintaining the position was recorded in seconds.

SECONDARY OUTCOMES:
instability | At baseline (pre-intervention) and 4 weeks after completing the intervention
  Ankle instability was assessed using the Cumberland Ankle Instability Tool (CAIT). The CAIT is a questionnaire developed to objectively evaluate symptoms of ankle instability. It consists of a total of 9 items, with a score range from 0 to 30. A score of 28 or higher indicates ankle stability, while a score of 24 or lower indicates ankle instability.
muscle strength | At baseline (pre-intervention) and 4 weeks after completing the intervention
  Ankle muscle strength was measured using a handheld dynamometer. Participants lay supine on a table, maintaining a straight position with the ankle and knee fully extended, and the ankle positioned at approximately 10-15° of plantar flexion at the edge of the table. Plantar flexion and dorsiflexion strength were measured by attaching the handheld dynamometer to the first metatarsal area. Each participant performed three trials of a 5-second maximal isometric contraction, with a 30-second rest between trials and a 90-second rest between sets. The assessor instructed participants to repeat a trial if maximal effort was not achieved or if posture was compromised.
function | At baseline (pre-intervention) and 4 weeks after completing the intervention
  Functional performance was assessed using the Side Hop Test. Participants stood on the unstable ankle and jumped side-to-side as quickly as possible between two parallel lines marked 30 cm apart. Each participant performed 10 consecutive jumps per set, completing a total of 3 sets with a 1-minute rest between sets. The test was considered complete when the participant successfully performed 10 jumps without stepping on the lines with the supporting foot or touching the ground with the non-supporting foot. The time to complete each set was recorded in seconds using a stopwatch, and the average time across the 3 sets was used for final analysis.

CONTACTS AND LOCATIONS:
Overall Officials: MIYONG JEONG, MSc, Principal Investigator — Sahmyook University Graduate School
Locations (1):
- Sahmyook University, Seoul, South Korea